CLINICAL TRIAL: NCT03342092
Title: Rebond d'adiposité précoce Chez l'Enfant de 4 Ans et Risque de Surpoids Chez l'Enfant de 11 Ans : troisième Temps d'Une Cohorte Franc-comtoise.
Brief Title: Early Adiposity Rebound Amongst 4-y.o. Children and Overweight Risk Amongst 11-y.o Children : Third Phase of a Cohort Study in Franche-Comté
Acronym: CoOP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2013/43
Record Dates: First submitted 2017-11-07; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Questionnaires distributed to the families 15 days before child's medical consultation
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires distributed to the families 15 days before child's medical consultation + anthropometric measures and data collected from the personal interview with school nurse

SUMMARY:
This study aims to assess different methods for early adiposity rebound determination at the age of 4/5 years old according to current medical screening criteria in schools, and to assess their prognostic value for obesity amongst 11 years old pre-adolescents according to the known risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls born between 1st July 2003 and 30th June 2004
* Attending school in Haute-Saône
* Enrolled in the 2008 cohort survey

Exclusion Criteria:

* Children whose parents refused to take part in this cohort study.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children initially enrolled in two successive surveys of build evolution and overweight determinants among a children cohort (both surveys representing the first time of the cohort), conducted in 2008.
Sampling Method: Non-Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Body mass index of 11 years old pre-adolescents | month 22
  Composite outcome based on height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Pasteur, MD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No